CLINICAL TRIAL: NCT05746676
Title: Clinical and Radiographic Evaluation of Insulin Versus Hyaluronic Acid in Management of Periodontal Defects
Brief Title: Insulin Versus Hyaluronic Acid in Management of Periodontal Defects
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Naglaa Elwakeel, professor, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P-ME-23-01
Record Dates: First submitted 2023-02-13; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Periodontal Diseases; Periodontal Pocket
Keywords: periodontitis; insulin; regeneration
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket; Periodontitis; Insulin Resistance | interventions — Insulin; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Active Comparator)
  Interventions: Drug: Insulin
- group 2 (Active Comparator)
  Interventions: Drug: Hyaluronic acid

INTERVENTIONS:
Drug: Insulin — in treatment of periodontal defects
  Arms: group 1
Drug: Hyaluronic acid — in treatment of periodontal defects
  Arms: group 2

SUMMARY:
in this study, insulin and hyaluronic acid will be used after open flap debridement in treatment of periodontal defects. outcome will be evaluated clinically and radiographically

DETAILED DESCRIPTION:
n this study, insulin versus hyaluronic acid will be used after open flap debridement in treatment of periodontal defects. outcome will be evaluated clinically and radiographically after a follow up period

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with periodontitis

Exclusion Criteria:

* patients with systemic illness that contraindicate periodontal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
clinical evaluation | 6 months
  periodontal pocket depth
radiographic evaluation | 6 months
  bone gain assessed by cone beam computed tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided